CLINICAL TRIAL: NCT06980428
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD4954 Following Single and Multiple Ascending Dose Administration to Healthy Participants With or Without Elevated Lp(a) Levels, and Participants With Dyslipidemia
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD4954 in Healthy Adult Participants With or Without Elevated Lipoprotein (a) (Lp[a]) Levels, and Participants With Dyslipidemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D7300C00001
Record Dates: First submitted 2025-05-19; First posted 2025-05-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Dyslipidemia
Keywords: Lipoprotein(a); Low-density lipoprotein cholesterol (LDL-C)
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Part A1: SAD Cohort 1 - AZD4954 (Dose 1) (Experimental): Participants will receive a single dose of AZD4954 (Dose 1) or matching placebo on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A1: SAD Cohort 2 - AZD4954 (Dose 2) (Experimental): Participants will receive a single dose of AZD4954 (Dose 2) or matching placebo on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A1: SAD Cohort 3 - AZD4954 (Dose 3) (Experimental): Participants will receive a single dose of AZD4954 (Dose 3) or matching placebo on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A1: SAD Cohort 4 - AZD4954 (Dose 4) (Experimental): Participants will receive a single dose of AZD4954 (Dose 4) or matching placebo on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A1: SAD Cohort 5 - AZD4954 (Dose 5) (Experimental): Participants will receive a single dose of AZD4954 (Dose 5) or matching placebo on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A1: SAD Optional Cohort 6 - AZD4954 (Dose 6) (Experimental): Participants will receive a single dose of AZD4954 (Dose 6) or matching placebo on Day 1. This additional cohort may be added depending on the findings.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A1: SAD Cohort 1 (Japanese) - AZD4954 (Dose 2) (Experimental): Japanese participants will receive a single dose of AZD4954 (Dose 2) or matching placebo on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A1: SAD Cohort 2 (Japanese) - AZD4954 (Dose 3) (Experimental): Japanese participants will receive a single dose of AZD4954 (Dose 3) or matching placebo on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A1: SAD Optional Cohort 3 (Japanese) - AZD4954 (Experimental): This additional cohort may be added depending on the findings.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A1: SAD Cohort 1 (Chinese) - AZD4954 (Dose 5) (Experimental): Chinese participants will receive a single dose of AZD4954 (Dose 5) or matching placebo at the highest dose level on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A2: SAD Food Effect Cohort - AZD4954 (Dose 2) (Experimental): Participants will receive a single dose of AZD4954 (Dose 2) or matching placebo with a high-calorie, high-fat breakfast on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part A2: SAD Food Effect Cohort - AZD4954 (Dose 3) (Experimental): Participants will receive a single dose of AZD4954 (Dose 3) or matching placebo with a high-calorie, high-fat breakfast on Day 1.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part B: Global MAD Cohort 1 (healthy participants) - AZD4954 (Dose 1) (Experimental): Participants will receive multiple doses of AZD4954 (Dose 1) or matching placebo for 21 days.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part B: Global MAD Cohort 2 (healthy participants) - AZD4954 (Dose 2) (Experimental): Participants will receive multiple doses of AZD4954 (Dose 2) or matching placebo for 21 days.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part B: Global MAD Cohort 3 (healthy participants) - AZD4954 (Dose 3) (Experimental): Participants will receive multiple doses of AZD4954 (Dose 3) or matching placebo for 21 days.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part B: Optional Global MAD Cohort 4 (healthy participants) - AZD4954 (Experimental): Participants will receive multiple doses of AZD4954 or matching placebo for 21 days. This additional cohort may be added depending on the findings.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part B: MAD Cohort (Japanese) - AZD4954 (Dose 3) (Experimental): Japanese participants will receive multiple doses of AZD4954 (Dose 3) or matching placebo for 21 days.
  Interventions: Drug: AZD4954; Drug: Placebo
- Part B: Global MAD Cohort (participants with dyslipidemia) - AZD4954 (Dose 1) (Experimental): Participants with dyslipidemia will receive multiple doses of AZD4954 (Dose 1) or matching placebo for 21 days.
  Interventions: Drug: AZD4954; Drug: Placebo

INTERVENTIONS:
Drug: AZD4954 — AZD4954 will be administered orally.
Drug: Placebo — Placebo will be administered orally.

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single and multiple ascending doses of AZD4954 in healthy participants with or without elevated Lipoprotein(a) (Lp[a]) levels and participants with dyslipidemia.

DETAILED DESCRIPTION:
This is a first time in human, placebo-controlled, single and multiple ascending dose (SAD and MAD) study in healthy male and female participants (Part A) or healthy participants with elevated Lp(a) levels (≥ 30 mg/dL) and participants with dyslipidemia with elevated Lp(a) levels (≥ 70 mg/dL) and low-density lipoprotein cholesterol (LDL-C) ≥ 70 mg/dL and < 190 mg/dL (Part B).

The study consists of 2 parts: Part A (SAD) and Part B (MAD).

Part A of the study will consist of Part A1 and Part A2, comprising:

* A Screening Period of maximum 28 days.
* Admission to study site (Day -1).
* A Treatment Period (Day 1 to Day 15 at the study site) with a single dose of AZD4954 or placebo on Day 1.
* A Follow-up Visit within 26 to 30 days after the study intervention dose for all cohorts (Day 29 ±2 days).

Part B has 3 types of MAD cohorts - global cohorts with healthy participants, global cohort with participants with dyslipidemia, and a Japanese cohort. The global MAD cohorts (healthy participants) and Japanese MAD cohort will comprise:

* A Screening Period of maximum 28 days.
* Admission to study site (Day -1).
* A Treatment Period during which participants will receive either AZD4954 or placebo once daily for 21 days (Day 1 to 21).
* A Follow-up Visit within 26 to 30 days after the last study intervention dose (Day 49 ±2 days).

The global MAD cohort (participants with dyslipidemia) will comprise:

* A Screening Period of maximum 28 days.
* Residential study site visits from Day -1 to Day 2 and Day 21 to Day 22.
* Non-residential study site visits on Day 8 and Day 15.
* A Treatment Period during which participants will receive either AZD4954 or placebo once daily for 21 days (Day 1 to 21).
* A Follow-up Visit within 26 to 30 days after the last study intervention dose (Day 49 ± 2 days).

ELIGIBILITY:
Inclusion Criteria:

All Parts:

* Participants with plasminogen level (concentration) within normal range at the Screening Visit.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the study site.
* Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception.
* Females of non-childbearing potential must be confirmed at the Screening Visit.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the study specific contraception methods from the time of first administration of study intervention until 3 months after the study Follow-up Visit.

Parts A and B (Healthy Participants):

* Male and female participants aged 18 to 65 years with suitable veins for cannulation or repeated venipuncture.
* Have a body mass index (BMI) between 18 and 35 kg/m² inclusive.
* For Japanese and Chinese participants (Parts A and B):

  1. A Japanese participant is defined as having both parents and 4 grandparents who are ethnically Japanese. This includes second and third generation Japanese whose parents or grandparents are living in a country other than Japan.
  2. A Chinese participant is defined as having both parents and 4 grandparents who are ethnically Chinese. This includes second and third generation Chinese whose parents or grandparents are living in a country other than China.

     Part B (Healthy Participants):
* Participants must have elevated Lp(a) ≥ 30 mg/dL at the Screening Visit.

Part B (Participants with Dyslipidemia):

* Male and female participants aged 18 to 70 years with suitable veins for cannulation or repeated venipuncture.
* Have a BMI > 18 kg/m².
* Participants must have elevated Lp(a) ≥ 70 mg/dL at the Screening Visit.
* Participants with a fasting LDL-C ≥ 70 mg/dL and < 190 mg/L at the Screening Visit.
* Participants should be receiving moderate or high-intensity statin therapy for ≥ 2 months prior to the Screening Visit, according to the American College of Cardiology/American Heart Association guidelines on blood cholesterol management.
* Participants with documented coronary artery disease, stroke, or peripheral artery disease or at moderate or high risk for an atherosclerotic cardiovascular disease event.
* There should be no planned medication or dose change during study participation.

Exclusion Criteria:

All Parts:

* History of any clinically important disease or disorder.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Participants with known bleeding or coagulation disorders.
* Participants who have an elevated high-sensitivity C-reactive protein (> 3 mg/L) or have a prothrombin time/international normalized ratio (PT/INR) or activated partial thromboplastin time (aPTT) > 1.25 times × upper limit normal (ULN).
* Any clinically important abnormalities in hematology, coagulation, clinical chemistry, urinalysis, abnormal vital signs or abnormal laboratory values.
* Any positive result on Screening for serum hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) or human immunodeficiency virus (HIV).
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead electrocardiogram (ECG) at Screening.
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of study intervention.

Parts A and B (Healthy Participants):

* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, intake of > 3 × daily recommended levels of vitamins and minerals during the 2 weeks prior to the first administration of study intervention or longer if the medication has a long half-life.
* Current smokers or those who have smoked or used nicotine products.

Part B (Participants with Dyslipidemia):

* Acute ischemic cardiovascular event in the last 12 months prior to randomization.
* Poorly controlled diabetes.
* Previous administration of Lp(a) inhibitor.
* Have uncontrolled hypertension.
* Abnormal vital heart rate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-12-04 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Screening (Day -28 to Day -2) to Follow-up visit (Up to Day 29±2 days)
  To assess the safety and tolerability of AZD4954 following oral administration of SAD (Part A).
Part B: Number of participants with AEs and SAEs | From Screening (Day -28 to Day -2) to Follow-up visit (Up to Day 49±2 days)
  To assess the safety and tolerability of AZD4954 following oral administration of MAD (Part B).

SECONDARY OUTCOMES:
Part A: Area under concentration-time curve from time 0 to infinity (AUCinf) | Up to Day 29±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Part B: Area under concentration-time curve in the dosing interval (AUCtau) | Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Dose normalized AUClast (AUClast/D) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Dose normalized AUCinf (AUCinf/D) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Part B: Dose normalized AUCtau (AUCtau/D) | Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Apparent total body clearance (CL/F) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Maximum observed drug concentration (Cmax) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Dose normalized Cmax (Cmax/D) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Terminal elimination half-life (t1/2λz) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Time of last quantifiable concentration (tlast) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Time to reach maximum observed concentration (tmax) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Apparent volume of distribution based on the terminal phase (Vz/F) | Part A: Up to Day 29±2 days; Part B: Up to Day 49±2 days
  To characterize the single dose and/or steady state pharmacokinetics of AZD4954 following oral administration of AZD4954.
Individual and cumulative amount of unchanged drug excreted into urine from time t1 to time t2 (Ae[t1-t2]) | Part A: Up to Day 15; Part B: Up to Day 22
  To characterize the single dose and/or steady state urine pharmacokinetics of AZD4954 following oral administration of AZD4954.
Cumulative amount of unchanged drug excreted into urine (Aeinf) | Part A: Up to Day 15; Part B: Up to Day 22
  To characterize the single dose and/or steady state urine pharmacokinetics of AZD4954 following oral administration of AZD4954.
Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 (fe[t1-t2]) | Part A: Up to Day 15; Part B: Up to Day 22
  To characterize the single dose and/or steady state urine pharmacokinetics of AZD4954 following oral administration of AZD4954.
Renal clearance (CLR) | Part A: Up to Day 15; Part B: Up to Day 22
  To characterize the single dose and/or steady state urine pharmacokinetics of AZD4954 following oral administration of AZD4954.
Part B: Absolute change from baseline in serum Lp(a) | Up to Day 49±2 days
  To evaluate the pharmacodynamics of AZD4954 by assessment of Lp(a) levels following repeated oral dosing.
Part B: Relative change from baseline in serum Lp(a) | Up to Day 49±2 days
  To evaluate the pharmacodynamics of AZD4954 by assessment of Lp(a) levels following repeated oral dosing.
Part B: Absolute change from baseline in Lp(a) intact assay | Up to Day 49±2 days
  To evaluate the pharmacodynamics of AZD4954 by assessment of Lp(a) levels following repeated oral dosing.
Part B: Relative change from baseline in Lp(a) intact assay | Up to Day 49±2 days
  To evaluate the pharmacodynamics of AZD4954 by assessment of Lp(a) levels following repeated oral dosing.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Glendale, California
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Brooklyn, Maryland
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/